## A Culturally Sensitive Intervention for TBI Caregivers in Latin America

PI: Paul Perrin, PhD

**NCT #**: 02207803

Virginia Commonwealth University Internal Review Board (IRB): HM20001660

Document approval date: 5/6/2014

**Document Type:** SAP

What is the TAP's impact on Latino caregivers' health status, burden, depression, sense of coherence, quality of informal care provided, and relationship satisfaction? Analytic Plan: A Greenhouse-Geisser-adjusted repeated measures multivariate analysis of variance (RMANOVA) with one fixed effect of treatment group (TAP vs. control), the repeated measures over time (baseline, and 2 and 4 months after discharge), and the treatment group by time interaction will be conducted for the set of dependent variables in Q1. If an omnibus effect is found, follow-up Bonferroni-corrected ANOVAs will identify specific locations of effects. These dependent variables rarely correlate with each other higher than .60,61 so do not reach the .70 level that Tabachnik and Fidell62 identify as problematic.

What is the TAP's impact on Latino TBI patients' functional and health status, self-perceived burden, depression, perceptions of quality of informal care received, and relationship satisfaction?

Analytic Plan: The same analyses will be used for the patient dependent variables.